CLINICAL TRIAL: NCT03597568
Title: Effect of 6 Weeks Resveratrol Supplementation on Vascular Function in CKD
Brief Title: Resveratrol and Vascular Function in CKD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diana Jalal (Other)
Responsible Party: Sponsor-Investigator, Diana Jalal, Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201806073
Record Dates: First submitted 2018-07-13; First posted 2018-07-24 (Actual); Results first posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-08

CONDITIONS: Chronic Kidney Diseases; Endothelial Dysfunction
Keywords: Resveratrol; Kidney Diseases; Renal Insufficiency; Diabetes; Oxidative stress; Endothelial dysfunction
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Diseases; Renal Insufficiency; Diabetes Mellitus | interventions — Resveratrol

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to either receive the following intervention: placebo or resveratrol for six weeks and then after a two week washout will be assigned the alternate study drug.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Resveratrol first, then placebo (Experimental): Patients will receive resveratrol 400 mg PO per day in divided doses of 200 mg in the morning and 200 mg in the evening. After a minimum of 2 week washout period, subjects then took placebo for 6 weeks.
  Interventions: Dietary Supplement: Resveratrol; Other: Placebo
- Placebo first, then resveratrol (Placebo Comparator): Patients will receive placebo pill identical in appearance and taste to the supplement. Subjects took this placebo twice daily, once in the morning and once in the evening. After a minimum of 2 week washout period, subjects then took resveratrol for 6 weeks.
  Interventions: Dietary Supplement: Resveratrol; Other: Placebo

INTERVENTIONS:
Dietary Supplement: Resveratrol — Oral supplementation for 6 weeks
Other: Placebo — Oral supplementation for 6 weeks

SUMMARY:
The proposed research is clinical study evaluating the therapeutic benefits of resveratrol on vascular function in patients with chronic kidney disease (CKD). The study aims to establish that resveratrol will improve endothelial function and functional performance by reducing oxidative stress and in conjunction with lowering markers of inflammation and oxidative stress.

DETAILED DESCRIPTION:
Patients with chronic kidney disease (CKD) have an exceptionally high risk for cardiovascular disease (CVD), and are 10 times more likely to die from CVD prior to requiring dialysis or kidney transplantation. Inflammation, oxidative stress and vascular dysfunction (impaired endothelial function and increased large elastic artery stiffness), are highly prevalent in CKD and contribute to the high incidence of CVD in this patient population. In addition, patients with CKD suffer from high rates of cognitive decline for which we lack effective therapies. Thus, therapeutic interventions targeting inflammation, oxidative stress, vascular dysfunction in CKD are a priority.

Wine intake, which is known to be rich in various polyphenolic compounds, might have a variety of health benefits. Among these polyphenols, the stilbene derivative resveratrol (RSV), a naturally occurring polyphenol found in grapes and red wine, has recently come to light, as it has been shown to exert potent anti-diabetic, anti-oxidative and anti-inflammatory actions. Importantly, recent studies have demonstrated that resveratrol is well-tolerated (37) and may confer similar benefits in individuals at high risk of CVD, such as improved endothelial function in individuals with metabolic syndrome (i.e. diabetes)

The primary goal of this application is to determine whether 6 wks resveratrol (RSV) supplementation improves vascular function by reducing oxidative stress in a randomized, double-blind, cross-over study of 25 patients with diabetic kidney disease. The investigators hypothesize that: 1) 6 wks RSV will improve vascular function as measured via BA-FMD vs. placebo and 2) that the improvement in vascular function will be related, at least partially, to a reduction in oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

* CKD stage III (estimated GFR: 30-60 mL/MIN/1.73m2)
* Able to give informed consent
* Angiotensin converting enzyme inhibitor or angiotensin II receptor bloocker for > 3 month prior to the study
* Type II diabetes mellitus

Exclusion Criteria:

* Consuming > 2 glasses/day red wine and/or taking resveratrol or vitamin C supplement in the past 12 months
* Life expectancy <1 year
* BMI >40 kg/m2 1
* Pregnant, breastfeeding, or unwilling to use adequate birth control
* Uncontrolled hypertension; blood pressure > 140/90
* Uncontrolled type II DM; AIC > 8.5
* Currently taking anticoagulants including: coumadin, dalteparin, enoxaparin, haparin, and plavix.
* Severe liver disease
* Severe systolic heart failure
* Hospitalization within the last 3 months
* Active infection or antibiotic therapy
* Immunosuppressive therapy within the last year
* Currently partaking in another research study

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-01-12 (Actual); Study Completion 2023-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diana Jalal, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gimblet CJ, Kruse NT, Geasland K, Michelson J, Sun M, Mandukhail SR, Wendt LH, Eyck PT, Pierce GL, Jalal DI. Effect of Resveratrol on Endothelial Function in Patients with CKD and Diabetes: A Randomized Controlled Trial. Clin J Am Soc Nephrol. 2024 Feb 1;19(2):161-168. doi: 10.2215/CJN.0000000000000337. Epub 2023 Oct 16. PMID 37843843

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Consented 28 and randomized 25
Pre-assignment Details: Randomized cross over design, each subject served as their own control. Randomized either to placebo first or resveratrol first. There was 2 week wash-out period.
Groups:
- Resveratrol First: Subjects received resveratrol 400 mg PO per day for 6 weeks then placebo after 2 week wash out period
- Placebo First: Subjects received placebo identical to the study drug for 6 weeks then resveratrol at 400 mg a day after a 2 week wash out
Period: Overall Study
Arm/Group | Resveratrol First | Placebo First
Started | 13 | 12
Completed | 11 | 10
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Unable to analyze vascular data | 1 | 1

BASELINE CHARACTERISTICS:
Population: Each subject functioned as their own control in this randomized cross over study
Groups:
- Resveratrol First; Placebo First: Randomized cross over design, subjects received either resveratrol or placebo first, 2 weeks washout separated the 2 treatments
- Total: Total of all reporting groups
Arm/Group | Resveratrol First | Placebo First | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Categorical [Count of Participants; unit: Participants] — Population: 2 subjects in total in both arms did not have vascular images that could be analyzed.
  Participants
    number analyzed (Participants) | 13 | 10 | 23
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 2 | 2 | 4
    >=65 years | 11 | 8 | 19
Age, Continuous [Mean (Full Range); unit: years] | 68 [50 to 74] | 69 [49 to 77] | 68 [49 to 77]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 2 subjects did not have vascular images that could be analyzed
  Participants
    number analyzed (Participants) | 13 | 10 | 23
    Female | 2 | 1 | 3
    Male | 11 | 9 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 2 subjects did not have vascular images that could be analyzed
  Participants
    number analyzed (Participants) | 13 | 10 | 23
    Hispanic or Latino | 0 | 0 | 0
    Not Hispanic or Latino | 13 | 10 | 23
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 2 subjects did not have vascular images that could be analyzed
  Participants
    number analyzed (Participants) | 13 | 10 | 23
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 13 | 10 | 23
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 10 | 23

OUTCOME MEASURES:

1. Primary Outcome: % Change of Brachial Artery Flow-mediated Dilation
Description: Brachial artery flow-mediated dilation, dilation of the brachial artery in response to shear stress.
  Resveratrol first, then placebo:
  Baseline to 6 weeks on Resveratrol Minimum 2 week washout Baseline to 6 week on placebo
  Placebo first, then resveratrol:
  Baseline to 6 weeks on placebo Minimum washout 2 weeks Baseline to 6 weeks on resveratrol
Time Frame: First Baseline measurement to 6 weeks then Second baseline to 6 weeks
Population: Randomized cross over design
Measure: Mean (95% Confidence Interval); unit: %change
Groups:
- Resveratrol: Resveratrol was compared to placebo in randomized cross over design
- Placebo: Randomized cross over design
Arm/Group | Resveratrol | Placebo
Number analyzed (Participants) | 21 | 21
%change | 1.3 [1.06 to 1.61] | 0.91 [0.74 to 1.12]

2. Secondary Outcome: Change in oxLDL
Description: Oxidized low density lipoprotein- (LDL) cholesterol Compare the 6 weeks change from baseline with resveratrol versus placebo
Time Frame: 6 weeks
Population: oxLDL was measured and change from baseline was compared for both groups.
Measure: Mean (95% Confidence Interval); unit: U/L
Groups:
- Resveratrol: This was compared to placebo, randomized cross over design
Arm/Group | Resveratrol | Placebo
Number analyzed (Participants) | 21 | 21
U/L | 1.66 [1.15 to 2.32] | 1.38 [0.98 to 1.94]

ADVERSE EVENTS:
Time Frame: 6 weeks of resveratrol supplementation
Groups:
- Resveratrol; Placebo: 6 weeks randomized cross over study, randomized to resveratrol first or placebo first, there was 2 week wash out period
Arm/Group | Resveratrol | Placebo
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 1/25 | 0/25
Other Adverse Events (participants affected / at risk) | 3/25 | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Resveratrol (N=25) | Placebo (N=25)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Subject reported dyspnea and admitted to hospital for supplemental oxygen.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Resveratrol (N=25) | Placebo (N=25)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0
Dizziness (General disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-23): https://cdn.clinicaltrials.gov/large-docs/68/NCT03597568/Prot_SAP_000.pdf